CLINICAL TRIAL: NCT02923037
Title: Feasibility and Preliminary Efficacy of Hatha Yoga in Breast Cancer Survivors: Pilot Study
Brief Title: Hatha Yoga in Breast Cancer Survivors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient staff and funding
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sheila Ridner, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VICC BRE 16104; NCI-2016-01402 (Registry Identifier: NCI, Clinical Trials Reporting Program)
Record Dates: First submitted 2016-09-29; First posted 2016-10-04 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Breast Carcinoma; Lymphedema
MeSH Terms: conditions — Breast Neoplasms; Lymphedema | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive Care (Yoga) (Experimental): Patients undergo an initial yoga evaluation for 60 minutes. Patients then undergo their first guided yoga practice session for 30-60 minutes and subsequent guided yoga sessions for 30-90 minutes 3 times a week for 4 weeks, and twice a week for an additional 4 weeks. Patients are also encouraged to complete home yoga practice for 30 to 90 minutes every day for 8 weeks. They will have tape measurement of arms and ldex measurement of arms. Quality-of-Life Assessment will also be made.
  Interventions: Procedure: Yoga; Other: tape measurement of arm; Other: Quality-of-Life Assessment; Other: ldex measurement of arms

INTERVENTIONS:
Procedure: Yoga — Complete guided and home yoga sessions
Other: tape measurement of arm — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies
Other: ldex measurement of arms

SUMMARY:
This pilot clinical trial studies Hatha yoga in reducing physical and emotional problems in breast cancer survivors with stage II-III lymphedema. Yoga practices may benefit breast cancer survivors with lymphedema as they directly support lymph transport (postures, breathing, relaxation) and emotional well-being (relaxation, meditation).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of a modified yoga program for breast cancer survivors (BCS) with lymphedema.

II. To identify and document required modifications for a safe and feasible practice.

III. To obtain recruitment estimates and determine barriers to recruitment (acceptability).

IV. To evaluate implementation fidelity (adherence and competence) and barriers to implementation fidelity.

V. To establish safety. VI. To assess satisfaction. VII. To determine the preliminary efficacy of a modified yoga program for lymphedema in BCS, and associated physical and psychological symptoms/symptom burden, and overall health status.

OUTLINE:

Patients undergo an initial yoga evaluation for 60 minutes. Patients then undergo their first guided yoga practice session for 30-60 minutes and subsequent guided yoga sessions for 30-90 minutes.

3 times a week for 4 weeks, and twice a week for an additional 4 weeks. Patients are also encouraged to complete home yoga practice for 30 to 90 minutes every day for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

Lymphedema Group:

* Lymphedema, symptomatic of stage II or III based upon screening responses; or L-Dex reading of ≥ 7 at initial visit,
* > 3 months (mths) post-breast cancer treatment
* No active cancer
* Has compression sleeve
* Ability to understand English in order to complete questionnaires
* Willing to do guided and home yoga practice
* Willing and able to provide informed consent as demonstrated by passing screening tool questions that includes the Short Portable Mental Status Questionnaire
* Medical clearance
* Reliable transportation to the study site

No Lymphedema Group:

* No known lymphedema or intermittent swelling, not symptomatic of Stage II or III lymphedema (L-Dex ≥ 7)
* >3 months post- breast cancer treatment
* No active cancer
* Ability to understand English in order to complete questionnaires
* Willing to do guided and home Yoga practice
* Willing and able to provide informed consent as demonstrated by passing screening tool questions that includes the Short Portable Mental Status Questionnaire
* Medical clearance
* Reliable transportation to the study site.

Exclusion Criteria (Both Groups):

* Active cancer
* Undergoing radiation therapy or chemotherapy
* Medical conditions that would prohibit the safe implementation of a yoga practice (e.g., vertigo, compromised mental status)
* Active yoga practice < 3 months
* Currently undergoing phase I complete decongestive therapy (CDT)
* Inability to complete study forms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Pose Modifications | Up to 8 weeks
  number of poses requiring modifications as indicated in the modification form
Assess safety | Up to 8 weeks
  Number of participants with treatment-related adverse events as assessed by the CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Ridner, PhD, RN, Principal Investigator — Vanderbilt University School of Nursing
Locations (1):
- Vanderbilt University School of Nursing, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided